CLINICAL TRIAL: NCT03180346
Title: A Prospective, Randomized, Comparative Study to Assess the Prevention of Surgical Site Infection (SSI's) in Revision Total Joint Arthroplasty Patients Treated With Single-Use Negative Pressure Wound Therapy (PICO) or Standard Care Dressings (AQUACEL Ag SURGICAL Dressing).
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 16Chen02
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Surgical Incision
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-Use Negative Pressure Wound Therapy (Active Comparator)
  Interventions: Device: PICO
- Standard of Care (Active Comparator)
  Interventions: Device: Aquacel

INTERVENTIONS:
Device: PICO — Single Use Negative Pressure Dressing
  Arms: Single-Use Negative Pressure Wound Therapy
Device: Aquacel — Occlusive surgical dressing infused with ionized silver
  Arms: Standard of Care

SUMMARY:
The primary aim of this study is to determine if the SSI rate following revision total hip and knee arthroplasty is reduced in patients treated with the PICO device compared to patients with traditional postoperative dressings. Our secondary goals include; comparing the amount of wound drainage, rate of resolution of wound drainage, length of hospital stay, functional outcomes, and economic implications of wound drainage and SSI after revision arthroplasty comparing PICO and traditional dressings.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥18 years old
2. Male or non-pregnant, non-lactating, postmenopausal or surgically sterilized females
3. Subjects undergoing revision total knee arthroplasty or revision total hip arthroplasty
4. Subjects provide informed consent, which will consist of reading, signing, and dating the informed consent document after the Investigator, sub-Investigator or other designated study staff member has explained the study procedures, risks, and contact information
5. Subjects deemed able to understand and comply with study visit schedule and procedures

Exclusion Criteria:

1. Wounds that require daily inspection
2. Active bleeding within the surgical site
3. Pregnant, lactating females, or females of childbearing potential not willing to practice an effective method of contraception
4. Subjects on warfarin therapy. Resulting in increased exudate and prolonging hospital stay following surgery to achieve therapeutic INR levels
5. Skin integrity issues that preclude the use of Negative Pressure Wound Therapy (NPWT)
6. Subjects undergoing primary total joint procedures
7. Subjects with a known history of poor compliance with medical treatment
8. Subjects who have participated in this trial previously and who were withdrawn 9 . Subjects with known allergies to product components (silicone adhesives and polyurethane films (direct contact with wound), acrylic adhesives (direct contact with skin), polyethylene fabrics and super-absorbent powders (polyacrylates) (within the dressing)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Estimated)
Dates: Start 2017-03-21 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection | 90-day followup following revision surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States